CLINICAL TRIAL: NCT03137680
Title: Effect Of Pre-Operative Forearm Exercise On Arteriovenous Fistula Mauration and Blood Flow
Brief Title: Pre-Operative Forearm Exercise On Arteriovenous Fistula Mauration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Sreekanth Koduri, Consultant, Changi General Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/2573
Record Dates: First submitted 2017-04-28; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Arteriovenous Fistula
Keywords: Arteriovenous Fistula; Pre-operative Exercise; Fistula Maturation
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Care Provider i.e., vascular surgeon are blinded to subject randomisation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): No specific exercise regime for the control group. Usual hospital SOP will be adhered to
- Exercise Arm (Experimental): The exercise protocol for the intervention group will be to squeeze a soft ball 10 times for set and perform 3 sets of 10 squeezes each at an 1 minute interval. Three sets of exercises to be performed twice in the morning and twice in the evening, for a total of 6 weeks. This will be performed at least 6 weeks prior to the creation of the AV fistula
  Interventions: Behavioral: Hand Exercise

INTERVENTIONS:
Behavioral: Hand Exercise — Exercise protocol for the intervention group will be to squeeze a soft ball 10 times for set and perform 3 sets of 10 squeezes each at an 1 minute interval. Three sets of exercises to be performed twice in the morning and twice in the evening, for a total of six weeks.
  Arms: Exercise Arm

SUMMARY:
To investigate the effect of pre-operative exercise on

1. Hemodynamics in the fistula artery and vein, pre and post AV fistula formation
2. Suitability of cannulation of AV fistula at 8weeks

DETAILED DESCRIPTION:
Aim: To investigate the effect of pre-operative exercise on hemodynamics in the fistula artery and vein, pre and post AV fistula formation as well as the suitability of cannulation of AV fistula at 8weeks post sugery

Methodology: This is a randomised control study with 20 patients each in the exercise arm and the control arm. The subjects will be randomised 1:1 into one of the two groups. Chronic Kidney failure patients with eGFR less than 20mls/min and have chosen Haemodialysis as their modality of renal replacement therapy will be included the study. All the subjects will have an ultrasound doppler vein mapping done prior to entering the study.

The exercise protocol for the intervention group will be to squeeze a soft ball 10 times for set and perform 3 sets of 10 squeezes each at an 1 minute interval. Three sets of exercises to be performed twice in the morning and twice in the evening, for a total of six weeks.

All patients will have a follow up ultrasound doppler of the AV fistula at 8 weeks and 16 weeks post-surgery, looking at the AV fistula vein diameter, arterial diameter and blood flow rate. All the subjects will also be seen by a single vascular surgeon following the scan, to assess the suitability for AVF cannulation.

Significance of the proposed study and benefits: A well functioning arterio-venous fistula is the gold standard vascular access for Hemodialysis patients due to its low rates of complications. The primary failure rate of the AVFs remain high at around 20 -25%, contributed by several factors including the diameter of the vessels. If pre-operative exercise improves the hemodynamics of the AV fistula and aids the maturation rate in our study, it can be incorporated into clinical guidelines to reduce the primary failure rate of AV fistulas.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic Kidney failure patients with eGFR less than 20mls/min
2. Chosen Hemodailysis as their modality of renal replacement therapy

Exclusion Criteria:

1. Potential fistula vein diameter less than 3mm (with application of tornique) on initial vein mapping
2. Known left ventricular ejection fraction of less than 20% on Echocardiogram
3. Previous stroke effecting the AV fistula arm
4. Calcified brachial or radial arteries and/or duplex evidence of stenosis of >50%

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2018-12-15 (Estimated); Study Completion 2019-03-20 (Estimated)

PRIMARY OUTCOMES:
Hemodynamics in the fistula artery and vein, pre and post AV fistula formation | 22 weeks
  AV fistula vein diameter, arterial diameter and blood flow rate will be assessed and compared

SECONDARY OUTCOMES:
Suitability of cannulation of AV fistula | 8 Weeks
  Assessment of suitability of AV fistula cannulation by blinded vascular surgeon 8 week post creation
Secondary fistula failure | 1 year
  Fistula outcomes will be assessed to review the need for angiographic procedures for AVF maturation and also look at secondary fistula failure

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nantakool S, Reanpang T, Prasannarong M, Pongtam S, Rerkasem K. Upper limb exercise for arteriovenous fistula maturation in people requiring permanent haemodialysis access. Cochrane Database Syst Rev. 2022 Oct 3;10(10):CD013327. doi: 10.1002/14651858.CD013327.pub2. PMID 36184076